CLINICAL TRIAL: NCT01266278
Title: Analysis of Sport Specific Adaptations of the Shoulder in Adolescent Elite Handball Players and the Influence of the Preventive Use of Tape on Shoulder Strength, Mobility, the Position of the Scapula and the Size of the Subacromial Space.
Brief Title: Analysis of Sport Specific Adaptations of the Shoulder in Adolescent Elite Handball Players and the Influence of the Preventive Use of Tape on These Outcome Measurements.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Prof. Dr. Ann Cools, University Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EC/2010/637
Record Dates: First submitted 2010-12-14; First posted 2010-12-24 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Risk Factors for Shoulder Injuries
Keywords: shoulder injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kinesiotape (Experimental): Kinesiotape will be applied to the correct shoulder position of the participants.
  Interventions: Other: Dynamic ultrasound; Other: FASTRAK; Other: Assessment of shoulder posture by measuring

INTERVENTIONS:
Other: Dynamic ultrasound — Measurement of the size of the subacromial space with dynamic ultrasound.
Other: FASTRAK — Measurements of the 3D-kinematics of the shoulder with FASTRAK. Sensors are placed on the skin of the shoulder with adhesive tape.
Other: Assessment of shoulder posture by measuring — Assessment of shoulder posture by measuring several angles and distances.

SUMMARY:
Shoulder complaints are very common in overhead athletes.The application of kinesiotape that keeps the shoulder in a correct position is used to avoid this.

This could enlarge the dynamic size of the subacromial space and thus contribute to prevention of shoulder injuries.

30 young elite handball players will participate in this study.Researchers will perform a number of measurements before and after applying kinesiotape to correct shoulder position:

* measurement of subacromial space
* measurement of 3D kinematics of shoulder
* assessment of shoulder posture

Hypothesis of this study is that tape can influence the position of the scapula and is therefore able to change the size of the subacromial space.This results in a more efficient use of shoulder muscles with higher maximal strength as a result and maximizes shoulder mobility.

DETAILED DESCRIPTION:
Shoulder complaints are very common in overhead athletes. Throwing motions question large explosive strength and stability of the intrinsic instable shoulder joint. Malpositioning of the scapula increases the risk of overload injuries.

The application of kinesiotape that keeps the shoulder in a correct position is used to avoid this. Until now no studies have shown if the tape is able to correct the position of the scapula. If this is the case, the application of the tape could enlarge the dynamic size of the subacromial space (virtual space in the shoulder in which rotator cuff tendons run through) and thus contribute to prevention of shoulder injuries.

This study will take place in collaboration with Prof. Dr. Robert Van Cingel, director of the Sports Medical Center Papendal(SMCP) in the Netherlands. SMCP is a multidisciplinary center for sports medicine, sports rehabilitation and sports cardiology.

30 young elite handball players will participate in this study. Three researchers will perform a number of measurements before and after applying kinesiotape to correct shoulder position.

1. Measurement of the size of the subacromial space with dynamic ultrasound. Ultrasound is completely harmless and painless.
2. Measurement of three-dimensional kinematics of the shoulder with FASTRAK. Sensors are placed on the skin of the shoulder with adhesive tape. Both placement of markers and measurements are non-invasive and painless.
3. Assessment of shoulder posture by measuring several angles and distances. Measurement of shoulder strength and mobility. These measurements are all non-invasive and painless.

Hypothesis of this study is that tape can influence the position of the scapula and is therefore able to change the size of the subacromial space. This results in a more efficient use of shoulder muscles with higher maximal strength as a result and maximizes shoulder mobility.

ELIGIBILITY:
Inclusion Criteria:

* Elite handball players of Papendal
* age between 15 and 25
* more than 15 hours of handball training/week
* female

Exclusion Criteria:

* shoulder pain at the moment for which a doctor was consulted

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
effect of kinesiotape | 2 days
  Immediate effects of applying kinesiotape to the correct shoulder position

CONTACTS AND LOCATIONS:
Overall Officials: Ann Cools, Ph.D., Principal Investigator — University Ghent
Locations (1):
- Sports Medical Center of Papendal, Arnhem, Netherlands